CLINICAL TRIAL: NCT07100847
Title: Phase 1b Window of Opportunity Study of Peri-prostatic Neurolysis in High-risk Localized Prostate Cancer
Brief Title: Periprostatic Neurolysis in Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Urology Care Foundation (Unknown); American Urological Association (Other)
Responsible Party: Principal Investigator, Ali Zahalka, Urologic Oncology Fellow, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU20240058
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: PROSTATE CANCER; NERVES; NEUROBIOLOGY OF CANCER; NEUROLYSIS
Keywords: HIGH RISK LOCALIZED PROSTATE CANCER
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single injection neurolysis (Experimental): Single injection of ethanol for periprostatic neurolysis
  Interventions: Procedure: Periprostatic neurolysis with dehydrated alcohol (ethanol)
- Two injection neurolysis (Experimental): Two temporally separated periprostatic ethanol injections
  Interventions: Procedure: Periprostatic neurolysis with dehydrated alcohol (ethanol)
- No injection control (No Intervention)

INTERVENTIONS:
Procedure: Periprostatic neurolysis with dehydrated alcohol (ethanol) — Pre-operative ultrasound guided periprostatic neurolysis by injection of dehydrated alcohol
  Arms: Single injection neurolysis; Two injection neurolysis

SUMMARY:
The purpose of this research study is to assess whether inhibiting nerve activity to the prostate delays progression of disease in men with high-risk clinical features for prostate cancer. Prostate cancer has been shown to invade nerves, a mechanism that is thought to be involved in prostate cancer spread in men with high-risk cancer. When nerve activity to the prostate is blocked in mice with prostate cancer, prostate cancer growth and spread are inhibited. In a previous study we showed that doing so in humans was safe and may have anticancer therapeutic effect. In this study we will test whether one versus two injections of nerve blocking agent is more effective at reducing nerves in the prostate and whether it will slow/stop spread of prostate cancer after treatment.

DETAILED DESCRIPTION:
Men with high-risk prostate cancer are at the greatest risk for clinical progression, with 22 to 40% developing metastatic disease within 10 years of initial treatment. Furthermore, the finding of perineural invasion (PNI) on pathology (when prostate cancer cells invade the nerves that innervate the prostate), is associated with higher Gleason grades and an approximate doubling in risk of lethal prostate cancer. As 90% of prostate cancer metastasis involve the bone marrow, and 97% of bone marrow metastasis involve the lumbar vertebrate from which the pre-ganglionic sympathetic nerves that innervate the prostate derive, targeting this neuro-anatomic connection between the prostate and its primary site of metastasis is an active area of investigation. Therefore, development of therapeutic strategies targeting nerves to prevent clinical progression after definitive therapy for prostate cancer are urgently needed. In a Phase 1a dose escalation study (NCT06703437) we recently demonstrated that periprostatic neurolysis with 5mL pure ethanol was well tolerated with no AEs. This resulted in an approximate 30% reduction in prostatic adrenergic nerve density. The goal of this study is to optimize prostatic denervation by comparing the denervation efficiency of 1 vs 2 periprostatic ethanol injections.

ELIGIBILITY:
Inclusion criteria:

High risk prostate cancer as defined by NCCN criteria Desires surgical disease treatment (radical prostatectomy) Surgical candidate (for radical prostatectomy)

≤cT3a on MRI No seminal vesicle, lymph node, or metastatic disease on PSMA PET No prior prostate cancer treatment (including androgen deprivation therapy, radiation therapy, focal therapy, cryo therapy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Peritumoral adrenergic nerve density on final histology | 4 to 6 weeks after treatment initiation
  Will quantify degree of neurolysis by measuring decrease in adrenergic nerve density on radical prostatectomy specimen histology

SECONDARY OUTCOMES:
Change in sexual health inventory for men (SHIM) score | 4 to 6 weeks after intervention
  Change in erectile function as measured by SHIM score at enrollment and 4 to 6 weeks after periprostatic neurolysis
Change in International Prostate Symptom Score (IPSS) | 4 to 6 weeks after intervention
  Change in lower urinary tract symptoms as measured by IPSS questionnaire at baseline and after neurolysis
Change in post prostatectomy penile length | 6months after surgery
  Change in penile length post prostatectomy compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.

REFERENCES:
- [Background] Zahalka AH, Arnal-Estape A, Maryanovich M, Nakahara F, Cruz CD, Finley LWS, Frenette PS. Adrenergic nerves activate an angio-metabolic switch in prostate cancer. Science. 2017 Oct 20;358(6361):321-326. doi: 10.1126/science.aah5072. PMID 29051371